CLINICAL TRIAL: NCT01737307
Title: Effect of Fluoride Varnish and CPP-ACP Paste on Oral and Salivary Symptoms of Patients Under Chemotherapy: A Double-blind Clinical Trial
Brief Title: Effect of Fluoride Varnish and CPP-ACP on Oral and Salivary Symptoms During Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sepideh Banava.DDS,MS, Assistant Professor Of Restorative Department, Azad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AZadUMS
Record Dates: First submitted 2012-11-15; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Mucositis; Dry Mouth; Infection
Keywords: Fluoride Varnish; CPP-ACP paste; Dry mouth; Burning sensation; Chemotherapy
MeSH Terms: conditions — Mucositis; Xerostomia; Infections; Paresthesia | interventions — Oral Hygiene; Toothbrushing; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fluoride Varnish (Experimental): Fluoride varnish was used once in this group. Fluoride varnish(NaF 5%,Sultan,USA)
  Interventions: Drug: Fluoride varnish
- Oral hygiene (Experimental): Oral hygiene followed twice daily. No F varnish or CPP-ACP applied.
  Interventions: Other: Oral Hygiene
- CPP-ACP (Experimental): CPP-ACP paste (GC Tooth Mousse,Gc,USA)was applied by patients once daily. 3gr,for 42 days.
  Interventions: Drug: CPP-ACP

INTERVENTIONS:
Drug: Fluoride varnish — Fluoride Varnish (NaF 5%)
  Other Names: Fluoride varnish(NaF 5%,Sultan,USA)
  Arms: Fluoride Varnish
Other: Oral Hygiene — Oral hygiene followed.
  Other Names: Twice daily (tooth brush and tooth paste).
  Arms: Oral hygiene
Drug: CPP-ACP — CPP-ACP paste was applied by patient, once daily.
  Other Names: CPP-ACP Paste was used in this group.; 3 gr , once daily , 42 days.
  Arms: CPP-ACP

SUMMARY:
The purpose of this study was to investigate the effect of Fluoride varnish and Casein Phospho-Peptide Amorphous Calcium Phosphate (CPP-ACP) containing paste on oral symptoms and salivary characteristics in patients under chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy as a treatment method of cancers, affects different parts of the oral cavity such as oral mucosa, teeth and salivary glands caused by salivary glands dysfunction during chemotherapy.Oral status of patients under chemotherapy will be affected by consumption of the drugs and their side effects such as reduction of the saliva, dryness of the oral cavity, changes in bacterial balance, oral mucosa damage, bleeding due to irritation of the tissues, xerostomia, dental caries, burning sensation, dysgeusia and dysphagia. No effective preventive protocol has been presented for oral care during chemotherapy.

Patients who were met the inclusion criteria (aged over 12, diagnosed to have cancer by an oncologists and needed chemotherapy drugs, had at least 20 teeth, had no other pathologic lesion in their oral cavity, were not treated by radiotherapy and did not have specific systemic diseases or head and neck cancer) were selected for the study. the participants were evaluated according to oral and salivary symptoms.

ELIGIBILITY:
Inclusion Criteria:

* to have cancer (in the first stage of their treatments)
* to have at least 20 teeth,
* age over 12

Exclusion Criteria:

* to have pathologic lesion in the oral cavity
* being under radiotherapy
* to have specific systemic diseases
* to have head and neck cancer

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
oral symptoms(mucositis, xerostomia, infection, dysphagia, dysgeusia, burning sensation in mouth. | 6 weeks after first visit

SECONDARY OUTCOMES:
pH of saliva | 6 weeks after first visit
pH of dental plaque | 6 weeks after first visit
Quantity of saliva ( rest and stimulated) | 6 weeks after first visit
Saliva buffering capacity | 6 weeks after first visit

CONTACTS AND LOCATIONS:
Overall Officials: Sepideh Banava, Assist-Prof, Principal Investigator — Azad University of Medical Sciences, Dental Branch
Locations (1):
- Azad University of Medical Sciences, Dental Branch, Tehran, Tehran Province, Iran